CLINICAL TRIAL: NCT01842555
Title: Photodynamic Therapy (PDT) Oncology Registry
Acronym: PDT Registry
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Main Line Health (Other)
Collaborators: Pinnacle Biologics Inc. (Industry)
Responsible Party: Principal Investigator, Patrick Ross, Principal Investigator, Main Line Health
Other Study IDs: R16-3560
Record Dates: First submitted 2013-04-18; First posted 2013-04-29 (Estimated); Last update posted 2018-08-24 (Actual); Status verified 2018-08

CONDITIONS: Lung Cancer; Esophageal
Keywords: PDT; Photodynamic therapy
MeSH Terms: conditions — Lung Neoplasms | interventions — Registries; 1-phenyl-3,3-dimethyltriazene

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- PDT registry patients: Any newly diagnosed lung or esophageal cancer that is being being treated with PDT at a participating institution.
  Interventions: Other: Registry

INTERVENTIONS:
Other: Registry — Registry
  Other Names: PDT

SUMMARY:
The data elements for the PDT Registry project include virtually all the elements in the standard hospital-based cancer registry record, although in some cases at a finer level of detail. All data points should be found in the participant's medical record. The principal difference between the PDT Registry data set and that collected by the registries is the inclusion of more information specific to PDT.

DETAILED DESCRIPTION:
Participating centers will need to describe its own mechanism for patient identification and eligibility screening. A data manager, identified by the Principal Investigator at each participating center, will screen all patients for eligibility. Appointment, diagnosis and treatment data will be reviewed using information such as clinic records, appointment lists, pathology department records, OR schedule and/or tumor registries. Patients meeting inclusion criteria will be enrolled in the 3-year registry which will comprise retrospective and prospective parts. Patients will be accrued retrospectively for the first 12-month period of the registry. The retrospective part will include patients who received PDT with Photofrin® from 2007 up to 2012. Patients who are eligible but die prior to enrollment will also be included to minimize bias resulting from non-inclusion of advanced stage patients. The prospective recruitment parts will be three years. The estimated length of follow-up for each patient will be 3 years. Follow-up will be conducted by research study staff at each institution via medical record review, under the direction of the Principal Investigator at that site. No patients will be contacted at any point to obtain study data or for follow-up.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older, male or female, diagnosed with cancer and is undergoing or has undergone Photodynamic Therapy (PDT).
* Patients must have undergone PDT with Photofrin® at a participating institution.
* Patients scheduled to undergo PDT with Photofrin®
* Cancer patients receiving some or all primary care (e.g.,cancer-directed surgery, systemic therapy, radiation therapy, palliative care)in the participating institution.
* Cancer patients with a history of any type of cancer who have been no evidence of disease(for five years but without a history of distant metastases or evidence of relapse if they meet the previous criteria).

Exclusion Criteria:

* Cancer patients who present to the participating institution with a diagnosis of a simultaneous second primary.
* Cancer patients receiving all primary cancer care (e.g., cancer-directed surgery, chemotherapy, targeted therapy, radiation therapy, palliative care) outside of participating institution.
* Patients treated with photosensitizers other than Photofrin®

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Each participating center will need to describe its own mechanism for patient identification and eligibility screening.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2012-11; Primary Completion 2024-11 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
A Photodynamic Therapy (PDT) research repository and de-identified registry | Up to 3 years
  Participating sites will be able to utilize aggregate, de-identified data to perform research on PDT, the patients receiving PDT, and their outcomes and complications after the procedure.
  Data collected includes the following:
  Table 1. Outline of Data Elements in the PDT Registry
  1. Patient Visit Form- Demographics Patient Identification Number Institution Number Study Type Surgeon ID Date of Birth Age at PDT Racial Background Gender Tobacco Use Alcohol Use Vital Status
  2. Pre-Treatment Primary Site Clinical Sta

SECONDARY OUTCOMES:
Survival following palliative and non-palliative PDT | Up to 3 years
  calculated by date of PDT treatment and date of death (where applicable)
Short and long term efficacy of PDT in presenting symptom improvement | Up to 3 years
  Quality of Life Score before and after PDT
Complications after PDT | up to 3 years after
  30-day mortality (yes/no), length of stay in hospital (number of days), assessment of PDT-related complications (ex: phototoxic reaction (yes/no), urgent re-bronchoscopy (yes/no))

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Ross, MD, PhD, Principal Investigator — Main Line Health
Locations (1):
- Main Line Health, Lankenau Medical Center, Wynnewood, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- See also: Main Line Healthcare System — http://www.mainlinehealth.org